CLINICAL TRIAL: NCT00544622
Title: Structured Stroke Management Improves Outcome at 6 Months
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kantonsspital Baden (Other)
Collaborators: 407 Doctors (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: INR50
Record Dates: First submitted 2007-10-12; First posted 2007-10-16 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-10

CONDITIONS: Stroke
Keywords: Stroke treatment; Rehabilitation; Stroke chain; Stroke unit
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: structured therapeutic chain of stroke treatment

SUMMARY:
Background/Aim of the study: To further reduce the 6 months stroke morbidity and mortality in a high volume stroke hospital and to compare the results with national and international data.

Methods: 204 consecutive stroke patients are analyzed in a prospective study in a single center teaching institution. The intervention consists of a structured therapeutic chain of 290 collaborating GPs, a standardised acute hospital proceeding overlapping with an early integrated neurovascular rehabilitation within the same institution. Primary endpoints include death and dependence at 6 months, secondary endpoints are the length of hospital stay (LOS) and the quantitative analysis of physical and psychosocial impairments. The data are directly compared with the same endpoints of the Swiss subgroup of the international stroke trial (IST).

ELIGIBILITY:
Inclusion Criteria:

* An acute cerebrovascular event (ischemic stroke or intra-cerebral bleeding (ICB)) with the signs and symptoms of an acute stroke according to the World Health Organisation definition of acute stroke14 within the last 12 hours without the need or possibility of a neurosurgical intervention
* No thrombolytic therapy within the first 3 hours (in order to allow the correct comparison with the Swiss cohort of the IST trial
* The informed consent of the patient or, if not possible, of the relatives
* Living at home before the event
* Lack of participation in another trial.

Exclusion Criteria:

* Thrombolytic therapy within the first 3 hours (in order to allow the correct comparison with the Swiss cohort of the IST trial
* No informed consent of the patient or, if not possible, of the relatives
* Not living at home before the event
* Participation in another trial (26 patients were excluded because of TIA with full recovery within 24 hours after the event)

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2002-01; Study Completion 2003-03

PRIMARY OUTCOMES:
Mortality, dependence, psychoscial outcome
Mortality, dependence and psychosocial outcome | 6 months endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Juerg H. Beer, MD, Study Chair — Department of Medicine

REFERENCES:
- [Derived] Langhorne P, Ramachandra S; Stroke Unit Trialists' Collaboration. Organised inpatient (stroke unit) care for stroke: network meta-analysis. Cochrane Database Syst Rev. 2020 Apr 23;4(4):CD000197. doi: 10.1002/14651858.CD000197.pub4. PMID 32324916